CLINICAL TRIAL: NCT06749080
Title: ASSIST 2.0: a Reablement Program for Healthy Ageing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aileen Bergström (Other)
Collaborators: Forte (Industry)
Responsible Party: Sponsor-Investigator, Aileen Bergström, PhD, Ass. Lecturer, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ASSIST 2.0
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Reablement; Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group - ASSIST intervention groups Uppsala/Stockholm (Active Comparator): All staff in the intervention group will recieve an on-line reablement education. The occupational and physcial therapist in the intervention group will provide mentoring including reflection for the homecare staff. Together the team will focus on the older persons everyday occuations and deliver reablement to the older persons.
  Interventions: Behavioral: Assist Reablement (including education and mentoring)
- Control group Uppsala/Stockholm (No Intervention): The older person will recieve home care as usual without a reablement education or support from occupational or physical therapists.

INTERVENTIONS:
Behavioral: Assist Reablement (including education and mentoring) — Reablement on-line education will be standard and mandatory for both intervention groups. Mentoring will be formed according to the pre-requisites at the site.
  Arms: Intervention group - ASSIST intervention groups Uppsala/Stockholm

SUMMARY:
The goal of this study is to continue to develop, implement, and evaluate a unique reablement service, ASSIST 2.0. The project will determine the differences in the reablement service (ASSIST 2.0) compared to regular home care in terms of older adults' performance in daily activities, self-efficacy, perceived health, quality of life, frailty and perceived person-centered approach.

The research question is: Can older adults receiving ASSIST 2.0 improve their performance and satisfaction in daily life activities, experience a higher level of self-efficacy, perceived health, quality of life and a person-centered approach?

The ASSIST project involves older adults receiving home care, home care assistants, occupational and physical therapists. ASSIST 2.0 reablement consists of the following components:

* an intervention aimed at older adults to help them perform daily activities they need and want to do. This will be achieved through optimal support from home care staff,
* an on-line education provided by the researchers for all staff in the art and science of reablement,
* training and support through mentorship and coaching provided by occupational and physical therapists for home care staff to ensure the proper delivery of reablement.

ELIGIBILITY:
Inclusion criteria:

* Homecare has been granted
* The person can describe an ordinary day and what they have problems with doing
* 65 years of age or over

Exclusion criteria:

• The person has palliative care

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
The improvement of performance and/or satisfaction in prioritized everyday activities after the end of the reablement intervention, 6 and 12 months post baseline. | Measurements will be at baseline, two weeks post base line, at the end of the intervention (6-12 weeks post baseline), 6 and 12 months post baseline.
  The Canadian Occupational Performance Measure (COPM) will be used. The COPM measures the level of self-assessed performanace and satisfaction of up to five prioritized everyday activities that the person needs, wants or is expected to do, but percieves difficulties doing them. The person rates, for each everyday activity, on a scale of 1 to 10 the prioritisation, the performance and the satisfaction of the activity. For the prioritisation 10 represents very important, one not important). For the performance scale, 10 represents the person does the activity extremely well, and one represents can not do the activity at all. For the satisfaction scale, 10 represents being extremely satisfied and and one not satisfied at all. An increase in two points or more from base-line to follow-up is a positive clinically significant difference.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Guidetti, PhD, Professor, Study Director — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Karolinska Institutet, Huddinge, Sweden
  - Uppsala Kommun, Uppsala, Sweden

REFERENCES:
- [Background] Assander S, Bergstrom A, Eriksson C, Meijer S, Guidetti S. ASSIST: a reablement program for older adults in Sweden - a feasibility study. BMC Geriatr. 2022 Jul 26;22(1):618. doi: 10.1186/s12877-022-03185-2. PMID 35879678